CLINICAL TRIAL: NCT00765752
Title: The Association of Cortical GABA Concentrations in Subjects With Primary Insomnia and Depression in Partial Remission With Residual Insomnia
Brief Title: Cortical GABA Concentrations in Insomnia
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Principal Investigator, Gerard Sanacora, Professor, Yale University
Other Study IDs: 0707002830; ESRC 057
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Insomnia; Major Depression
Keywords: Insomnia; depression; GABA; magnetic resonance spectroscopy; MRS; Sleep; antidepressant medication use
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 Primary Insomnia: Individuals with insomnia not related to another identified cause.
- 3 Healthy comparison subjects: Healthy subjects with no history of insomnia

SUMMARY:
Disturbances in the amino acid neurotransmitter (AANt), gamma-amino butyric acid (GABA) function are hypothesized to contribute to the neurobiology of Major Depressive Disorder (MDD) and insomnia. The principal objective of this project is to use magnetic resonance spectroscopy (MRS) to provide the first in vivo characterization of cortical GABA levels in individuals with primary insomnia, and to determine whether subjects with MDD, achieving a partial response with selective serotonin reuptake inhibitor treatment but still experiencing significant residual symptoms including insomnia, have altered levels of this neurotransmitter. The investigators are also exploring the correlation between cortical AANt levels and abnormalities in sleep parameters in primary insomnia and as a residual symptom of major depression.

DETAILED DESCRIPTION:
Three groups of subjects (MDD with partial remission and residual insomnia, primary insomnia, and healthy) will participate in the study. All subjects will complete a telephone screening, and if appropriate a complete face-to-face evaluation, to determine their eligibility for the study. All subjects meeting eligibility criteria for the study will complete a baseline MRS session to evaluate differences in GABA concentrations between the three groups.

ELIGIBILITY:
Patient Sample.

* Healthy subjects without insomnia (Group A) (n=10)
* Subjects with primary insomnia (Group B) (n=20)
* Subjects with a history of major depressive disorder and currently in partial remission but with residual insomnia (Group C) (n=20)

Inclusion Criteria for Primary Insomnia Subjects:

* Males or females between the ages of 25 and 55 years
* Clinical diagnosis of primary insomnia meeting DSM-IV criteria.
* Current insomnia ratings (current Sleep Onset Latency SOL > 30 minutes, Insomnia Severity Index (ISI) > 14, total sleep time (TST) < 6.5 hrs/night).
* No lifetime history of psychopathology other than primary insomnia.
* No sleep disorders previously identified as related to other conditions including sleep disordered breathing, restless leg syndrome, periodic limb movement disorder, chronic pain, gastro-esophageal reflux disease, sleep paralysis, nocturnal seizures, nocturia, enuresis; also narcolepsy and REM behavior disorders (assessed by clinical interview and Harvard Center and Cognition Habitual Sleep Survey).

Inclusion Criteria for Depressed Subjects:

* Males or females between the ages of 25 and 55 years
* Clinical diagnosis of major depression meeting DSM-IV criteria in partial remission (HDRS-8-17), confirmed after semi-structured interview with the SCID and HDRS.
* On monotherapy with a single SSRI medication for a period of at least 6-weeks.
* Remaining symptoms of insomnia (current Sleep Onset Latency (SOL) > 30 minutes, Insomnia Severity Index (ISI) > 14, TST < 6.5 hrs/night).
* Participation is judged clinically appropriate by treatment team.
* No sleep disorders previously identified as related to other conditions including sleep disordered breathing, restless leg syndrome, periodic limb movement disorder, chronic pain, gastro-esophageal reflux disease, sleep paralysis, nocturnal seizures, nocturia, enuresis; also narcolepsy and REM behavior disorders.

Inclusion Criteria for Healthy Control Subjects:

* Males or females between the ages of 25 and 55 years
* No lifetime history of psychopathology or insomnia (current SOL < 30mins, ISI < 4, TST > 6.5 hrs)
* At low risk for depression (e.g., no first degree relative with child onset, recurrent, psychotic or bipolar depression)

Exclusion Criteria for all Subjects:

* History of serious medical or neurological illness
* Signs of major medical or neurological illness on examination or as a result of laboratory studies
* History of psychoactive substance and/or alcohol dependence or abuse in past 6-months.
* Current use of any psychoactive medication or substance (with the exception of caffeine, as noted below, and the use of an SSRI in the depressed group), during the two weeks prior to the initial scan.
* More than the caffeine-equivalent of 3 cups of coffee per day, or any regular (i.e., more than 1x/2 weeks) use of caffeine after 7pm.
* Use of benzodiazepines or olanzapine in past 3-months.
* Pregnant or nursing
* Any implanted metal devise or metal fragments

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2007-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Cortical GABA levels as measured by proton MRS | baseline

SECONDARY OUTCOMES:
Ambulatory polysomnography | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Sanacora, M.D.,Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale Depression Research Program, New Haven, Connecticut, United States